CLINICAL TRIAL: NCT00664482
Title: A Single-Patient Study Using AGS 006 as an Immunotherapeutic in a Subject With Newly Diagnosed Resectable Pancreatic Cancer
Brief Title: A Single-Patient Study Using AGS 006
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-006-001
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AGS-006
  Interventions: Biological: AGS-006

INTERVENTIONS:
Biological: AGS-006 — Autologous Therapy for Pancreatic Cancer

SUMMARY:
Argos Therapeutics, Inc., (Argos) proposes to study AGS-006 in a subject with newly diagnosed resectable pancreatic cancer. The AGS 006 immunotherapeutic may potentially offer a desired additional option to conventional treatments for pancreatic carcinoma.

DETAILED DESCRIPTION:
Single-patient, open-label clinical study:

* Events during Pre-Treatment Period:

  1. Resection of pancreatic cancer,
  2. RNA acquisition from tumor specimen,
  3. RNA amplification,
  4. Infectious disease testing,
  5. Autoimmune disease testing,
  6. Two blood draws for immune response monitoring,
  7. Production leukapheresis, and
  8. Dendritic cell electroporation with RNA and immunotherapeutic production;
* Events during Induction Period:

  1. Administer investigative treatment every 2 weeks for a total of five doses, followed by dosing every 4 weeks for a total of four doses,
  2. Two Induction Period blood draws (Week 6 and Week 12) for immune response monitoring, and
  3. One leukapheresis (Week 14) for immune response monitoring;
* Events during Booster Period:

  1. Dose every 3 months until progression or 2 years after first AGS treatment,
  2. Potentially, one leukapheresis for immune response monitoring 12 months from the first dose, and
  3. One blood draw 2 weeks following dosing at Week 36 (1st booster dose) (approximately Week 38); and,
* Events during study Close-Out:

  1. Close-Out upon progression or 28 days following immune response monitoring 2 years after first dose

ELIGIBILITY:
Inclusion Criteria:

* A male subject 18 years of age or older with newly diagnosed resectable pancreatic cancer who, in the opinion of the investigator, is suitable for participation in the study will be eligible for inclusion if all of the following criteria apply:

  1. Able to abstain from taking prohibited prescription or prohibited non-prescription drugs.
  2. Ability to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the Protocol requirements.
  3. Voluntary informed consent given to participate in the study.

Exclusion Criteria:

1. Any serious medical condition such as cardiopulmonary disease, circulatory compromise, hepatic or renal dysfunction, or other illness considered by the investigator to constitute an unwarranted high risk for investigational treatment.
2. Active autoimmune disease including, but not limited to:
3. Active, acute, or chronic clinically significant infections including human immunodeficiency virus (HIV) and viral hepatitis.
4. Known hypersensitivity to dimethyl sulfoxide (DMSO).
5. Body weight less than 30 kg.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent changes in vital signs (blood pressure, heart rate, respiratory rate, and body temperature) from baseline values obtained prior to each investigative treatment
Incidence of treatment-emergent adverse events graded according to the Common Terminology Criteria for Adverse Events
Treatment-emergent adenopathy, tenderness, or inflammation (inguinal and axillary) assessed before and after each dose
Treatment-emergent changes in autoimmunity evaluations as measured by clinical signs and symptoms and laboratory assessments at periodic intervals during the Treatment Period.
Treatment-emergent changes in localized injection site reactions following each dose

SECONDARY OUTCOMES:
Assessment of progression-free survival (PFS) estimated from the date of subject registration - Standard Response Evaluation Criteria in Solid Tumors (RECIST) definitions of progressive disease (PD) will contribute to estimating the interval for PFS.
T cell response to RNA-electroporated DCs will be assessed by flow cytometry using blood cells collected according to protocol time and events
Positive immune response
Feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Schlesinger, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States